CLINICAL TRIAL: NCT00571597
Title: Prospective Analysis of the Wolf Minimaze Procedure for Treatment of Atrial Fibrillation
Brief Title: Short Term Outcomes From Minimally Invasive Surgery for the Treatment of Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM10695
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Atrial Fibrillation
Keywords: surgery; ablation; radiofrequency; minimaze; transtelephonic monitoring
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the efficacy of minimally invasive surgery for atrial fibrillation.

DETAILED DESCRIPTION:
Patients who are undergoing or who have undergone minimally invasive surgery for atrial fibrillation will be followed prospectively. At 6 to 9 months, 1 and two years post surgery follow-up subjects will receive a trans-telephonic monitor to wear for approximately 1 month, and will submit transmissions on a daily basis. Episodes of atrial fibrillation will be documented during this time. The overall efficacy of the procedure will be assessed based on the freedom from atrial fibrillation at the time of transtelephonic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* paroxysmal, persistent, or permanent atrial fibrillation

Exclusion Criteria:

* concomitant heart surgery requiring open thoracotomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be male or females age 18-85 that have elected to undergo or have undergone a minimally invasive "minimaze" surgery for the treatment of atrial firillation
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2007-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Transtelephonic monitoring for the identification of post surgical Atrial Fibrillation | six months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Ellenbogen, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Division of Cardiology Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Han FT, Kasirajan V, Kowalski M, Kiser R, Wolfe L, Kalahasty G, Shepard RK, Wood MA, Ellenbogen KA. Results of a minimally invasive surgical pulmonary vein isolation and ganglionic plexi ablation for atrial fibrillation: single-center experience with 12-month follow-up. Circ Arrhythm Electrophysiol. 2009 Aug;2(4):370-7. doi: 10.1161/CIRCEP.109.854828. Epub 2009 Jun 2. PMID 19808492
- [Background] Han FT, Kasirajan V, Wood MA, Ellenbogen KA. Minimally invasive surgical atrial fibrillation ablation: patient selection and results. Heart Rhythm. 2009 Dec;6(12 Suppl):S71-6. doi: 10.1016/j.hrthm.2009.07.027. Epub 2009 Oct 24. PMID 19864190
- [Result] Kasirajan V, Spradlin EA, Mormando TE, Medina AE, Ovadia P, Schwartzman DS, Gaines TE, Mumtaz MA, Downing SW, Ellenbogen KA. Minimally invasive surgery using bipolar radiofrequency energy is effective treatment for refractory atrial fibrillation. Ann Thorac Surg. 2012 May;93(5):1456-61. doi: 10.1016/j.athoracsur.2012.01.110. PMID 22541178